CLINICAL TRIAL: NCT03968861
Title: Neurological Outcome After 24 Months of Age Following Treatment With Xenon Combined With Moderate Hypothermia After Perinatal Asphyxia
Brief Title: Outcome After 24 Months of Participants in the TOBY Xenon Study
Status: Completed | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS157755
Record Dates: First submitted 2019-05-14; First posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Perinatal Asphyxia; Encephalopathy
MeSH Terms: conditions — Brain Diseases | interventions — Xenon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard care with moderate hypothermia: Surviving children allocated to standard care with moderate hypothermia in the TOBY-Xe trial
- 30% Xenon for 24 hours combined with moderate hypothermia: Surviving children allocated to inhaled xenon combined with moderate hypothermia in the TOBY-Xe trial
  Interventions: Drug: Xenon

INTERVENTIONS:
Drug: Xenon — Inhaled xenon gas given via purposely designed ventilator
  Other Names: Lenoxe
  Groups: 30% Xenon for 24 hours combined with moderate hypothermia

SUMMARY:
The objective of this study is to document the outcome at 2-3 years of age of participants of the TOBY Xe trial, to provide preliminary information about the later clinical effects of treatment with Xenon gas combined with moderate hypothermia following perinatal asphyxia. The TOBY Xe trial was a randomised controlled trial of inhaled xenon gas combined with hypothermia for the treatment of perinatal asphyxia. The trial primary outcome was changes on magnetic resonance parameters examined prior to discharge from hospital.

Continuing clinical follow-up of trial participants is important following any therapeutic trial and is essential in early phase trials where information on the clinical effects of the intervention are lacking. Therefore, we have set up this study to determine the major clinical and neurological outcomes of participants of the TOBY Xe trial and to determine whether the magnetic resonance parameters in that trial are qualified to predict outcome following neural rescue therapy. This information is necessary for planning further studies of this intervention.

ELIGIBILITY:
Inclusion Criteria:

Surviving participants in the TOBY Xenon study

Exclusion Criteria:

Lack of consent to participate

Ages: 2 Years to 3 Years | Sex: All
Age Groups: Child
Study Population: The study population were the surviving participants in the TOBY Xenon study. There were 69 survivors from 92 participants at 2 years after birth and 62 of the 69 participants entered the TOBY Xenon Follow-up Study
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Scores on Bayley scales of infant and toddler development | at 2-3 years of age
  Composite scores of the Cognitive, Language and Motor scales scaled to a metric, with a mean of 100, standard deviation of 15, and range of 40 to 160
Relation between magnetic resonance markers and neurodevelopmental outcome | at 2-3 years of age
  Peak area Lactate/N Acetyl Aspartate ratio on magnetic resonance spectroscopy and fractional anisotropy on diffusion tensor magnetic resonance imaging

SECONDARY OUTCOMES:
Grade of disability | At 2-3 years of age
  The grade of disability, categorised as mild disability (a Cognitive score of 70 to 84, level 1 gross motor function [is able to walk independently but may have some gait abnormalities], or abnormality in one or both eyes with normal or nearly normal vision), moderate disability (a Cognitive scale score of 56 to 69, level 2 or 3 gross motor function [has minimal ability to perform gross motor skills or requires assistance with walking], or moderately reduced vision), or severe disability (a Cognitive scale score of 55 (the minimum score on the Bayley Cognitive scale), level 4 or 5 gross motor function [needs adaptive seating or has severely limited mobility], or no useful vision).

OTHER OUTCOMES:
Optimality Scores on Hammersmith neurological examination | At 2-3 years of age
  Range of score is 0-78 with lower scores indicating more abnormal examination
Gross Motor Function Classification System | At 2-3 years of age
  Levels 1-5 with higher levels indicating worse neuromotor function
Manual Ability Classification System | At 2-3 years of age
  Levels 1-5 with higher levels indicating increasing difficulty in handling objects
Clinical signs of cerebral palsy | At 2-3 years of age
  Defined according to Surveillance of Cerebral Palsy in Europe classification.

CONTACTS AND LOCATIONS:
Overall Officials: David A Edwards, FMedSci, Principal Investigator — King's College London
Locations (3):
- United Kingdom (3):
  - Guys and St Thomas NHS Trust, London
  - Imperial College London NHS Healthcare Trust, London
  - University College London Hospital NHS Foundation Trust, London